CLINICAL TRIAL: NCT05324657
Title: Anatomical and Perioperative Predisposing Factor for Limb Occlusion of Incraft Infrarenal Endograft (LIMIT Study)
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, Principal Investigator, IRCCS San Raffaele
Other Study IDs: LIMIT Study
Record Dates: First submitted 2022-04-06; First posted 2022-04-12 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Aneurysm Abdominal
Keywords: abdominal aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim was to determine, within the patient enrolled in three controlled prospective studies, INNOVATION, INSPIRATION and INSIGHT (Sponsor: Cordis, A Cardinal Health Company) studies which are preoperative and postoperative anatomical risk factors associated to limb occlusion. In the three studies the total number of enrolled patients was 400, of whom 134 enrolled in the US

ELIGIBILITY:
Inclusion Criteria:

* Patients with abdominal aortic aneurysm, who have been treated with the INCRAFT® Grafting System (AAA Stent-Graft System).
* All cases treated with Incraft who were enrolled in three controlled prospective studies, INNOVATION, INSPIRATION and INSIGHT (Sponsor: Cordis, A Cardinal Health Company)

Exclusion Criteria:

* no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases treated with Incraft who were enrolled in three controlled prospective studies, INNOVATION, INSPIRATION and INSIGHT (Sponsor: Cordis, A Cardinal Health Company).
  The patients will be compared in order to detect possible significant differences in terms of perioperative risk factors that could affect the study. Risk adjustment or other statistical tools might be used to create comparable cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
limb occlusion | 30 days
  freedom from limb occlusion
freedom from death | 30 days
  survival

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Bruin JL, Baas AF, Buth J, Prinssen M, Verhoeven EL, Cuypers PW, van Sambeek MR, Balm R, Grobbee DE, Blankensteijn JD; DREAM Study Group. Long-term outcome of open or endovascular repair of abdominal aortic aneurysm. N Engl J Med. 2010 May 20;362(20):1881-9. doi: 10.1056/NEJMoa0909499. PMID 20484396
- [Background] United Kingdom EVAR Trial Investigators; Greenhalgh RM, Brown LC, Powell JT, Thompson SG, Epstein D, Sculpher MJ. Endovascular versus open repair of abdominal aortic aneurysm. N Engl J Med. 2010 May 20;362(20):1863-71. doi: 10.1056/NEJMoa0909305. Epub 2010 Apr 11. PMID 20382983